CLINICAL TRIAL: NCT02751645
Title: The Efficacy and Safety of Acute Normovolemic Hemodilution in Pediatric Cardiac Surgery Patients
Brief Title: Safety and Efficacy of Acute Normovolemic Hemodilution in Pediatric Cardiac Surgery Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Oregon Health and Science University (Other)
Collaborators: The Gerber Foundation (Other)
Responsible Party: Principal Investigator, Weronika Crescini, MD, Assistant Professor, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB#: 11949
Record Dates: First submitted 2016-04-13; First posted 2016-04-26 (Estimated); Last update posted 2019-05-16 (Actual); Status verified 2019-05

CONDITIONS: Cardiac Defect
Keywords: Pediatric; Cardiac; Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard of Care Control (No Intervention): This group will consist of all the participants that receive the standard of care treatment for elective surgical repair or palliation of their cardiac defect with the use of the cardiopulmonary bypass machine.
- Acute Normovolemic Hemodilution (Experimental): This group will consist of all the participants that receive the acute normovolemic hemodilution prior to their elective surgical repair or palliation of their cardiac defect with the use of the cardiopulmonary bypass machine.
  Interventions: Procedure: Acute Normovolemic hemodilution

INTERVENTIONS:
Procedure: Acute Normovolemic hemodilution — ANH is a technique in which a portion of the patients' own blood is removed before any surgical bleeding occurs. It is stored until the end of the operation, at which point it is returned to the patient.
  Arms: Acute Normovolemic Hemodilution

SUMMARY:
The investigators primary objective is to determine if acute normovolemic hemodilution (ANH) for pediatric cardiac surgical patients decreases the volume of blood products transfused during surgery and the immediate post-operative period as compared to usual care. This study will enroll 24 pediatric heart surgery patients, aged 6 months to 3 years old undergoing either ANH prior to initiating cardiopulmonary bypass or the standard of care procedures for the use of cardiopulmonary bypass.

DETAILED DESCRIPTION:
Blood transfusion has been associated with worse outcomes in pediatric cardiac surgical patients. The major complications associated with it include increased blood loss during and after surgery, kidney disease requiring dialysis, abnormal coagulation profile, increased vasopressor use, and increased time spent on the ventilator and in the intensive care unit. One strategy to minimize blood product administration is acute normovolemic hemodilution (ANH). The investigators primary aim is to determine if ANH for pediatric cardiac surgical patients decreases the volume of blood products transfused during surgery and the immediate post-operative period, compared to usual care. The investigators designed a randomized, controlled, open label study that equally assigns 24 pediatric cardiac surgery patients aged 6 months to 3 years into two groups to receive either ANH prior to initiating cardiopulmonary bypass or usual standard of care. Participants in the ANH arm of the study will have 10 ml/kg of blood removed following anesthetic induction. In order to maintain normal circulating volume, the collected blood will be replaced with an equal volume of 5% albumin. All participants will be treated with a standardized protocol aimed at blood conservation including the use of retrograde arterial and antegrade venous perfusion, small circuit size, intraoperative red blood cell salvage, and low hemoglobin targets to trigger transfusion.

ELIGIBILITY:
Inclusion Criteria:

* Informed signed consent must be obtained by a legally authorized representative.
* Must be undergoing an elective surgical repair or palliation of a cardiac defect with the use of the cardiopulmonary bypass machine.
* Must be clinically stable at the time of evaluation for eligibility and on the day of randomization.

Exclusion Criteria:

* Patients who carry a diagnosis of a bleeding disorder.
* Patients who have an abnormal coagulation profile as evidenced by a preoperative coagulation screen.
* Patients who have received a blood transfusion in the preceding 120 days.
* Patients who have a diagnosis of a chromosomal abnormality.
* Patients whose participation in the study is deemed unsafe by their primary care team.

Ages: 6 Months to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2016-06-30 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-05-31 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of ANH to decrease volume of blood products during surgery and the immediate post-operative period. | 2 Days
  This will be measured by comparing the volume (mL/Kg body weight) of any blood products administered peri-operatively between the two groups.

SECONDARY OUTCOMES:
Kidney function | 2 days
  This will be measured by the change in creatinine on postoperative day 2 from the pre-operative baseline value
Normalization of thromboelastogrpahy (TEG) MA value (maximum amplitude) | 2 days
  This will be measured by thromboelastography (TEG) test following end of cardiopulmonary bypass
Normalization of thromboelastography (TEG) R value (reaction time) | 2 days
  This will be measured by thromboelastography (TEG) test following end of cardiopulmonary bypass
Normalization of thromboelastography (TEG) Alpha Angle value | 2 days
  This will be measured by thromboelastography (TEG) test following end of cardiopulmonary bypass
Final hematocrit, platelet count, PT/PTT on ICU admission | 1 day
  These lab values will be recorded and compared for each group.
Hematocrit and platelet count on post-operative day 1 | 1 days
  These lab values will be recorded and compared for each group.
Time to end of vasoactive support in the first 24 hours post-operation. | 1 days
  This value will be recorded and compared for each group.
Duration of mechanical ventilation and ICU stay | 8 days
  This value will be recorded and compared for each group.

CONTACTS AND LOCATIONS:
Overall Officials: Miriam Treggiari, MD, Study Director — Oregon Health and Science University
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No
There are no plans to share the data collected during this study.